CLINICAL TRIAL: NCT03360370
Title: Screening for Neurodevelopmental Disorders in Children With Congenital Heart Disease Aged From 6 to 66 Months in Nord-Pas-de-Calais
Brief Title: Neurodevelopmental Disorders in Children With Congenital Heart Disease
Acronym: NeuroDis-CHD
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_31; 2017-A01839-44. (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Congenital Heart Disease
Keywords: Neurodevelopmental disorders,; Congenital heart disease; Children
MeSH Terms: conditions — Heart Defects, Congenital; Neurodevelopmental Disorders | interventions — Glycation End Products, Advanced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 6 to 66 months children with significant CHD: Children with "significant" congenital heart disease (CHD) aged from 6 to 66 months at the time of the study and fulfilling inclusion criteria for whom an age-appropriate questionnaire completed by parents (Ages & Stages Questionnaires, Third Edition in French (ASQ-3™) will be used to screen developmental delays.
  Interventions: Other: Ages & Stages Questionnaires, Third Edition in French (ASQ-3™)

INTERVENTIONS:
Other: Ages & Stages Questionnaires, Third Edition in French (ASQ-3™) — This questionnaire screens 5 neurodevelopmental areas (communication, gross motor, fine motor, problem solving and personal-social); 30 items per questionnaire about the child's abilities are evaluated.
  It takes about 15-20 minutes. Data are collecting and a scoring by a professional is provided. Follow-up action is taken for children at risk. Medical and surgical history is also collected to detect risk factors for neurodevelopmental disorders among neonatal data, characteristics of congenital heart disease and first surgery, and other comorbidities.

SUMMARY:
Children with congenital heart disease are at risk for neurodevelopmental disorders, these disorders impacting their quality of life and their integration into society.

The aim of this study is to detect neurodevelopmental disorders in children (aged from 6 to 66 months) with congenital heart disease in Nord-Pas-De-Calais (France) and to evaluate the frequency and risk factors of these neurodevelopmental disorders for a better follow-up.

This study will help implementing a specific program for the evaluation and management of neurodevelopmental disorders in children suffering from congenital heart disease in Nord-Pas-De-Calais and more globally, in the region Hauts-De-France.

DETAILED DESCRIPTION:
Are selected children with "significant" congenital heart disease (aged from 6 to 66 months) in "Nord-Pas-De-Calais" fulfilling inclusion criteria. A reliable and valid questionnaire used to screen developmental delays of children aged from one month to 66 months is completed by volunteer parents at the time of the study. Data of the questionnaire is collected and a scoring by professional is provided ; children at risk for neurodevelopmental delays are depicted.

In parallel, medical and surgical history is also collected to detect risk factors for neurodevelopmental disorders.

The frequency of neurodevelopmental disorders in this screened population according to risk factors (among neonatal data, severity of congenital heart disease, surgery, length of stay at hospital,... ) will be evaluated. The ratio children with neurodevelopmental disorders for whom specific care was implemented/ children with neurodevelopmental disorders who did not have specific care despite neurodevelopmental disorders will be established.

Follow-up action will be taken for children at risk for developping neurological disorders highlighted by the screening.

This study will help implementing a specific program for evaluation and management of neurodevelopmental disorders for children with congenital heart disease in our region.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 66 months at the time of study
* living in region "Nord-Pas-De-Calais"
* with " significant" congenital heart disease (= complex congenital heart diseases operated or not, simple or moderate congenital heart disease who had cardiac surgery)
* Followed by the Pediatric Cardiology Department of Lille University Hospital, or patients having a cardiopediatric follow-up outside Lille University Hospital but having been taken in charge at the University Hospital of Lille for any reason (cardiac or not)

Exclusion Criteria:

Children :

* lost to sight
* Deceased
* with congenital heart disease, living in Nord-Pas-de-Calais but never having been taken in charge at Lille University Hospital
* with mild or moderate congenital heart disease not having undergone surgery or having only undergone cardiac catheterization
* with cardiac surgery not performed in the Centers of Jacques CARTIER and Marie LANNNELONGUE

Ages: 6 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children With Congenital Heart Disease
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Percentage of children classified "at risk" for neuro-developmental disorders by the Age & Stage Questionnaire Third Edition in French (ASQ3) score | Baseline: one session
  The ASQ3 evaluates neurodevelopment in children by a parental questionnaire. ASQ-3 score screens 5 neurodevelopmental areas (communication, gross motor, fine motor, problem solving and personal-social); 30 items per questionnaire about the child's skills are evaluated. Each item could be range between Yes (The child do the action - 10 points), Sometimes (5 points) or Not yet (0 point). The scale for each areas could be from 0 (worse outcome) to 60 points (best outcome). The different areas scores are referred in a chart specific of each questionnaire. In each area the score indicates if the child's development appears to be on schedule (best outcome), need learning and attention or need to be evaluated by a professional (worse outcome, - 2 SD from the global population).

SECONDARY OUTCOMES:
Frequency of neurodevelopmental disorders in children with congenital heart disease in this screened population | Baseline: one session
  Number of children depicted with neurodevelopmental delays in comparison to children who do not have neurodevelopmental delays in the screened population
Frequency of neurodevelopmental disorders according to the severity of congenital heart disease | Baseline: one session
  Children with neurodevelopmental disorders are classified according to the severity of the congenital heart disease ( mild, moderate or severe congenital heart disease). The percentage of children with neurodevelopmental disorders in each category is established and compared to the others.
Number of Children With Documented Risk Factors for neurodevelopmental disorders | Baseline: one session
  The number of children with documented risk factors for neurodevelopmental disorders among neonatal data characteristics of congenital heart disease and first surgery, and comorbidities is evaluated
Ratio of children with neurodevelopmental disorders and for whom specific care was implemented | Baseline: one session
  The ratio of children with neurodevelopmental disorders for whom specific care was implemented /children with neurodevelopmental disorders who do not have specific care despite neurodevelopmental disorders is established

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Paule GUILLAUME, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, CHU, Lille, France

REFERENCES:
- [Derived] Billotte M, Deken V, Joriot S, Vaksmann G, Richard A, Bouzguenda I, Godart F, Baudelet JB, Rakza T, Nguyen The Tich S, Guillaume MP. Screening for neurodevelopmental disorders in children with congenital heart disease. Eur J Pediatr. 2021 Apr;180(4):1157-1167. doi: 10.1007/s00431-020-03850-x. Epub 2020 Oct 29. PMID 33119792